CLINICAL TRIAL: NCT03487432
Title: A ComparIson of Strategies to Prepare Severely Calcified Coronary Lesions - A Prospective Randomized Controlled Trial of Super High-Pressure NC PTCA Balloon Versus Scoring PTCA Balloon in Severely Calcified Coronary Lesions
Brief Title: A ComparIson of Strategies to PrepAre SeveRely CALCified Coronary Lesions
Acronym: ISAR-CALC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: SIS Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE Nr. BA00117
Record Dates: First submitted 2018-03-23; First posted 2018-04-04 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Calcified Coronary Artery Disease (Grade 3)
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPN NC (Experimental): Patients receiving a Super High-Pressure NC PTCA Balloon (OPN NC)
  Interventions: Device: Super High-Pressure NC PTCA Balloon (OPN NC)
- NSE Alpha (Experimental): Patients receiving a Scoring PTCA Balloon (NSE Alpha)
  Interventions: Device: Scoring PTCA Balloon (NSE Alpha)

INTERVENTIONS:
Device: Super High-Pressure NC PTCA Balloon (OPN NC) — Strategy of Super High-Pressure NC PTCA Balloon (OPN NC) after unsuccessful lesion preparation with conventional NC balloon angioplasty.
  Arms: OPN NC
Device: Scoring PTCA Balloon (NSE Alpha) — Strategy of Scoring PTCA Balloon (NSE Alpha) after unsuccessful lesion preparation with conventional NC balloon angioplasty.
  Arms: NSE Alpha

SUMMARY:
The objective of this prospective, multicenter, randomized, open-label trial is to evaluate the completeness of stent expansion following a strategy of lesion preparation with either a Super High-Pressure NC PTCA Balloon (OPN NC) or a Scoring PTCA Balloon (NSE Alpha) after unsuccessful lesion preparation with conventional NC balloon angioplasty in an angiographically well-defined group of patients with severely calcified coronary lesions (grade 3) undergoing coronary stent implantation (SYNERGY everolimus-eluting stent (EES)).

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years and consentable;
* Persistent angina symptoms despite optimal medical therapy and/or evidence of inducible ischemia;
* Angiographically-proven coronary artery disease;
* De novo lesion in a native coronary artery;
* Target reference vessel diameter between 2.25 and 4.00 mm by visual estimation;
* Calcification of the target lesion as determined by angiography (grade 3);
* Unsuccessful lesion preparation (<30% reduction of baseline diameter stenosis) with conventional NC balloon angioplasty
* Written informed consent.

Exclusion Criteria:

* Myocardial infarction (within 1 week);
* Limited long-term prognosis due to other conditions;
* Target lesion is in a coronary artery bypass graft;
* Target lesion is an in-stent restenosis;
* Target lesion is aorto-ostial;
* Target vessel thrombus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Stent expansion index (SEI) | intraprocedural
  Stent expansion index (SEI), defined as minimum stent area divided by mean reference area in an optical coherence tomography (OCT) quantitative analysis

SECONDARY OUTCOMES:
Angiographic Success | intraprocedural
  'Angiographic Success', defined as the achievement of residual angiographic stenosis <30% of the target lesion in the presence of TIMI 3 flow
Procedural Success | 30 days
  'Procedural Success', defined as the achievement of angiographic success without any MACE, defined as cardiac death, target vessel related myocardial infarction and repeat revascularization (PTCA/PCI or coronary artery bypass graft [CABG])
Strategy Success | intraprocedural
  'Strategy Success' defined as procedural success using the assigned study device and stent, without requirement for lesion preparations with further devices (i.e. rotational atherectomy [RA])
Acute lumen gain, | intraprocedural
  Acute lumen gain, defined as minimal lumen diameter (MLD) post balloon angioplasty minus baseline MLD (mm)
Complementary lesion preparations | intraprocedural
  Number of complementary lesion preparations with further devices (i.e. rotational atherectomy [RA])
Rate of vessel perforation | intraprocedural
  Rate of vessel perforation
Procedure duration | intraprocedural
  Procedure duration in min
Contrast volume | intraprocedural
  Contrast volume in mL

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Byrne, MD BCh PhD, Study Chair — Deutsches Herzzentrum Muenchen; Salvatore Cassese, MD PhD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (5):
- Germany (4):
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Herzzentrum Leipzig, Leipzig
  - Deutsches Herzzentrum Muenchen, München
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No